CLINICAL TRIAL: NCT03066245
Title: Autologous Bone Tissue Constructed On Biodegradable Polymer for the Treatment of Aneurysmal Bone Cysts
Brief Title: Use of Stem Cells Cultured on a Scaffold for the Treatment of Aneurysmal Bone Cysts (ABC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sophia Al-Adwan (Other)
Responsible Party: Sponsor-Investigator, Sophia Al-Adwan, Researcher, Msc, University of Jordan
Organization: University of Jordan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABCUJCTC
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Aneurysmal Bone Cyst
Keywords: Aneurysmal bone cysts; PLGA; Platelet Lysate; Bone marrow; Mesenchymal stem cells
MeSH Terms: conditions — Bone Cysts, Aneurysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC-PLGA (Experimental): The lesion will be treated with curettage then 1 million of bone marrow derived MSC seeded on 5x5 mm2 PLGA scaffold will be engrafted in the cyst of ABC patient.
  Interventions: Biological: MSC-PLGA

INTERVENTIONS:
Biological: MSC-PLGA — Bone marrow derived MSC seeded on biodegradable PLGA, supplemented with PL.

SUMMARY:
Patients qualified for this study are those diagnosed with ABCs and failed to be treated with other forms of classical therapies. In which, these patients will be engrafted with biodegradable scaffolds seeded with Mesenchymal Stem Cells (MSCs) supplemented with Platelet lysate.

DETAILED DESCRIPTION:
Aneurysmal bone cysts (ABC) are relatively rare, benign, tumor-like, expansile osteolytic lesions of unknown etiology which are predominantly found within the long bones and characterized by frequent idiopathic fractures. Despite the large variety of bone substitutes that have been used to fill these cystic lesions, to date there is no graft material which can be regarded as completely satisfactory, with a recurrence rate that ranges from 5-40% of treated cases. Autologous bone marrow derived mononuclear cells have been used previously to treat ABCs. Poly lactic-co-glycolic acid (PLGA) scaffolds have been used in bone tissue engineering due to their biodegradability and biocompatibility. Human platelet lysate (PL) contains a number of mitogenic growth factors and has been demonstrated to enhance mesenchymal stem cell (MSC) proliferation and expansion rate in vitro. This study is designed to assess the safety and effectiveness of using PLGA scaffolds seeded with autologous bone marrow MSCs and supplemented with osteogenic media and platelet lysate in healing bone lesions of patients suffering from aneurysmal bone cysts. This study will be conducted at the Cell Therapy Center (CTC), Jordan. Four ABC cases will be included. Patients qualified for this study are those diagnosed with ABCs and failed to be treated with other forms of classical therapies; such as allografts or who are not candidate of autografts.

ELIGIBILITY:
Inclusion Criteria:

* Bone cyst diagnosed with MRI, CT-scan, or X-Ray
* Intact cyst wall with high risk for fracture
* Cysts with minimum diameter of 6mm
* Diagnostic test performed on cyst fluid
* Diagnosed ABC patients whom treatments with other forms of classical therapies ;such as allograft failed or who are not candidate of autografts
* Provided written consent form

Exclusion Criteria:

* Patients with diagnosis of cancer
* Patients enrolled in other clinical trial

Ages: 4 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) as a result of the MSC-PLGA engraftment | 3 months
  The safety of the engraftment will be monitored by assessing any adverse event resulting from the engraftment procedure

SECONDARY OUTCOMES:
Effectiveness of using PLGA scaffolds seeded with autologous bone marrow MSCs by Radiograph | 6 months
  Patients will be followed up radiographically to evaluate bone filling at the site of the ABC

CONTACTS AND LOCATIONS:
Overall Officials: Abdalla Awidi, Study Director — University of Jordan
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided